CLINICAL TRIAL: NCT06886737
Title: Home-based Treatment of Binocular Eye Dysfunction in Veterans With Traumatic Brain Injury
Brief Title: Home-based Vision Therapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: N5317-R
Record Dates: First submitted 2025-03-07; First posted 2025-03-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Convergence Insufficiency
Keywords: Vision, Binocular; Convergence, Ocular
MeSH Terms: conditions — Ocular Motility Disorders

STUDY DESIGN:
Intervention Model Description: Participants perform convergence exercises at home in the form of a custom virtual-reality game. The trial is divided into two 6-week blocks, one for active treatment and one for no treatment. Participants will be randomized into the treatment-first or treatment-second arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Intervention block followed by non-intervention block
  Interventions: Other: Virtual-reality convergence training game
- Group B (Experimental): Non-intervention block followed by intervention block
  Interventions: Other: Virtual-reality convergence training game

INTERVENTIONS:
Other: Virtual-reality convergence training game — The participant plays a custom virtual-reality game that is designed to train convergence.

SUMMARY:
Post-concussive vision symptoms affect many Veterans who have experienced traumatic brain injury (TBI). One common issue is trouble with near vision, a problem that may persist long after the acute injury. Double vision or difficulty focusing on close objects can affect reading and depth perception. Poor reading can interfere with academic or work performance, and loss of near focusing can affect jobs that require fine motor tasks like machining and electrical work. Even having trouble using a smartphone can have a substantial impact on both work and social function. Near vision impairment after TBI is not well understood, and treatments are limited. The goal of this project is to investigate novel virtual-reality assessments and training games to improve the near vision diagnosis and home-based rehabilitation. Restoring normal near vision function could have a large impact on the fulfillment of Veterans' educational, career, and overall life goals.

ELIGIBILITY:
Inclusion Criteria:

* U.S. Military Veteran
* Place of residence within driving distance of Cleveland, OH
* Clinical eye exam within 6 months prior to enrollment and since the most recent TBI (if applicable) and the onset of near vision symptoms (if applicable)
* Best-corrected visual acuity 20/25 or better in each eye
* Convergence insufficiency (VR-NPC < 32 deg)

Exclusion Criteria:

* Neurological condition other than TBI that would affect convergence
* History of strabismus, amblyopia, or other binocular vision issues prior to TBI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-01-14 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Vergence Capacity (VR-NPC) | At study onset, At completion of Block 1 (six weeks duration), At completion of Block 2 (six weeks duration)
  The near point of convergence (angle of maximum ocular convergence) will be measured using a custom virtual-reality application.
System Usability Scale (SUS) | At completion of active treatment block (six-weeks duration)
  This is a standardized questionnaire to assess how easy a new technology is to use.
Simulator Sickness Questionnaire (SSQ) | At completion of active treatment block (six-weeks duration)
  This is a standardized questionnaire to test the player's tolerance of the virtual-reality experience.

SECONDARY OUTCOMES:
Accommodation | At study onset, At completion of Block 1 (six weeks duration), At completion of Block 2 (six weeks duration)
  Ocular accommodation (focus of the intraocular lens for near viewing) will be measured using the minus-lens method.
Dynamic Vergence | At study onset, At completion of Block 1 (six weeks duration), At completion of Block 2 (six weeks duration)
  The accuracy and speed of fixation steps between virtual near and far targets is assessed.
Stereoacuity | At study onset, At completion of Block 1 (six weeks duration), At completion of Block 2 (six weeks duration)
  Stereovision is assessed in virtual reality. Stereoacuity threshold is determined from a curve fit to the response data.
VR Word Reading: Word Accuracy Score | At study onset, At completion of Block 1 (six weeks duration), At completion of Block 2 (six weeks duration)
  The accuracy and speed of word reading is assessed in response to lists of words presented to the participant in virtual reality. The Word Accuracy Score is the number of words read correctly minus errors.
VR Word Reading: Reading Speed Score | At study onset, At completion of Block 1 (six weeks duration), At completion of Block 2 (six weeks duration)
  The accuracy and speed of word reading is assessed in response to lists of words presented to the participant in virtual reality. The Reading Speed Score is the Word Accuracy Score divided by total reading time.
WIAT Word Reading Tests: Word Accuracy Score | At study onset, At completion of Block 2 (six weeks duration)
  Participants read lists of words and nonsense words. The number of words read correctly is the accuracy score. Raw score will be converted to a standardized score (mean=100, S.D.=15) using normative data.
WIAT Word Reading Test: Word Fluency Score | At study onset, At completion of Block 2 (six weeks duration)
  Participant reads lists of words and nonsense words. The number of words read correctly within 30 seconds is the fluency score. Raw score will be converted to a standardized score (mean=100, S.D.=15) using normative data.
WIAT Oral Reading Fluency and Comprehension Test: Oral Reading Accuracy Score | At study onset, At completion of Block 2 (six weeks duration)
  Participant reads two passages aloud. The Oral Reading Accuracy Score is the number of words read minus errors (mispronunciations or additions). Raw score will be converted to a standardized score (mean=100, S.D.=15) using normative data.
WIAT Oral Reading Fluency and Comprehension Test: Oral Reading Fluency Score | At study onset, At completion of Block 2 (six weeks duration)
  Participant reads two passages aloud. The Oral Reading Fluency Score is the Oral Reading Accuracy Score (Outcome #9) divided by the time needed to complete reading of the passage. Raw score will be converted to a standardized score (mean=100, S.D.=15) using normative data.
Convergence Insufficiency Symptom Survey (CISS) | At study onset, At completion of Block 1 (six weeks duration), At completion of Block 2 (six weeks duration)
  This is a standardized questionnaire to assess symptoms related to near vision.

CONTACTS AND LOCATIONS:
Overall Officials: Mark F. Walker, MD, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No